CLINICAL TRIAL: NCT01213693
Title: Long-term Effects of Inhaled Corticosteroids (ICS) Treatment on Sputum Bacterial and Viral Loads in Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Effects of Inhaled Corticosteroids on Sputum Bacterial Load in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Alberto Papi, MD, Professor in Respiratory Medicine, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LTEICSBV01
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Bacteria; Virus; Inhaled Corticosteroids
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Virus Diseases | interventions — Fluticasone-Salmeterol Drug Combination; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICS/LABA group (Experimental): Patients assigned to this arm will take bid 50/500 mcg fluticasone/salmeterol combination
  Interventions: Drug: Salmeterol/Fluticasone combination
- LABA group (Active Comparator): Patients assigned to this arm will take bid 50 mcg salmeterol
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: Salmeterol/Fluticasone combination — Salmeterol/Fluticasone 50/500 mcg 1 inhalation bid
  Arms: ICS/LABA group
Drug: Salmeterol — Salmeterol 50 mcg 1 inhalation bid
  Arms: LABA group

SUMMARY:
Exacerbations are important events in the natural history of chronic obstructive pulmonary disease (COPD). Beside the acute (and prolonged) clinical impact, there is evidence that exacerbations negatively affect the natural history of the disease; e.g. lung function decline is accelerated in patients with frequent exacerbations. Bacteria are considered the most relevant cause of exacerbations, but there is evidence that viral infections are equally contributing.

Either alone or in combination with viruses, airway bacterial load in stable COPD correlates with both the frequency of exacerbations and the decline in lung function.

A long-term clinical trial recently showed that the regular treatment with inhaled corticosteroids (ICS) increases the risk of infectious events such as pneumonia, whereas it reduces the frequency of acute COPD exacerbations in COPD.

In a recent study it was found that airway bacterial load increases over time (1 yr follow up) in stable COPD. In this study, virtually all patients (93%) were treated with ICS.

This study is designed to evaluate whether long-term (1 year) ICS treatment increases viral and/or bacterial load in the sputum of COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Sixty stable moderate COPD patients (Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage 2) requiring regular treatment with long-acting bronchodilators, according to international guidelines.
* GOLD stage 2 COPD patients will be enrolled providing they were steroid-free for the last 4 months

Exclusion Criteria:

* Atopy
* Asthma
* Concomitant lung diseases (e.g. lung cancer)
* Acute infections of the respiratory tree in the previous 3 months including COPD exacerbation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
comparison between groups of bacterial load in sputum | 1 year
  The primary outcome will measure changes in sputum bacterial load of COPD patients treated with inhaled corticosteroids in combination with long acting beta-2 bronchodilators (ICS/LABA group) compared with COPD treated only with long acting beta-2 bronchodilators (LABA group)

SECONDARY OUTCOMES:
Correlations between clinical outcomes and sputum viral and/or bacterial load | 1 year
  To evaluate whether sputum viral and/or bacterial load correlate with symptoms and need for rescue medication in stabile COPD.
Sputum viral and/or bacterial load and exacerbation rate | 1 year
  To evaluate whether changes in sputum viral and/or bacterial load (end of the study vs baseline) correlate with exacerbation rate in COPD patients
Sputum viral and/or bacterial load and lung function | 1 year
  To evaluate correlations between changes in sputum viral and/or bacterial load and changes in lung function over 1 year.
Airway inflammation and viral/bacterial load in COPD | 1 year
  To evaluate correlations between sputum inflammatory cell profiles and markers of airway inflammation (interleukin-6) and viral/bacterial load at stable stable conditions in COPD paetints.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Papi, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Research Centre on Asthma and COPD - Department of Clinical and Experimental Medicine - Section of Respiratory Disease - University of Ferrara, Ferrara, Italy

REFERENCES:
- [Derived] Contoli M, Pauletti A, Rossi MR, Spanevello A, Casolari P, Marcellini A, Forini G, Gnesini G, Marku B, Barnes N, Rizzi A, Curradi G, Caramori G, Morelli P, Papi A. Long-term effects of inhaled corticosteroids on sputum bacterial and viral loads in COPD. Eur Respir J. 2017 Oct 5;50(4):1700451. doi: 10.1183/13993003.00451-2017. Print 2017 Oct. PMID 28982774